CLINICAL TRIAL: NCT03551067
Title: The Efficacy OF Oral DexmedetomidineVersus Oral Midazolam/Ketamine ON Parental Separation AND Face Mask Acceptance IN Pediatrics Undergoing Adenotonsillectomy
Brief Title: Oral Dexmedetomidine for Parental Separation in Pediatrics Undergoing Adenotonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mohamed A Elsadany, MD, Lecturer in Anesthesiology, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2886
Record Dates: First submitted 2018-05-08; First posted 2018-06-11 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Adenotonsillectomy
Keywords: Dexmedetomidine; Adenotonsillectomy; Parental Separation; Face Mask Acceptance
MeSH Terms: interventions — Dexmedetomidine; Adrenergic alpha-2 Receptor Agonists; Midazolam; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Patients received Dexmedetomidine (4 µg/kg) mixed with apple juice to fill the syringe up to 10 ml given orally once.
  Interventions: Drug: Dexmedetomidine
- Midazolam/Ketamine (Active Comparator): Patients received Midazolam (0.5 mg/kg) and Ketamine (1 mg/kg) mixed with apple juice to fill the syringe up to 10 ml given orally once.
  Interventions: Combination Product: Midazolam/Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine mixed with juice was given to the child orally preoperatively.
  Other Names: Alpha 2 agonist
  Arms: Dexmedetomidine
Combination Product: Midazolam/Ketamine — Midazolam/Ketamine was mixed with juice and given to the child orally preoperatively
  Other Names: Dormicum/Katalar
  Arms: Midazolam/Ketamine

SUMMARY:
The efficacy of oral dexmedetomidine as sedative versus a combination of oral midazolam plus oral ketamine were compared regarding to satisfactory separation from parents, satisfactory mask induction and postoperative rescue analgesia in Pediatrics undergone Adenotosillectomy

DETAILED DESCRIPTION:
After obtaining approval from the research Ethics Committee of the Suez Canal University Hospitals and written informed consent from the parents of each participant, 74 American Society of Anesthesiologists (ASA) physical status I and ІІ children aged 3-10 years scheduled for adenotonsillectomy under general anesthesia were enrolled into the study.

Patients were randomly assigned into one of two equal groups on alternative basis using closed envelope method; 37 patients for each group.

Group (D): Patients who received oral dexmedetomidine (4 µg/kg) mixed with apple juice to fill the syringe up to 10 ml.

Group (MK): Patients who received a combination of oral midazolam (0.5 mg/kg) and oral ketamine (1 mg/kg) mixed with apple juice to fill the syringe up to 10 ml.

Methods:

I- Preoperative visit:

During the preoperative visit, the following was done:

1. A written informed consent from the parents of each participant was obtained.
2. The techniques were explained to the parents including benefits and complications.

II- Preoperative assessment:

This includes:

A) Medical history:

1. Medical disorders (as diabetes, heart, chest, liver or kidney diseases).
2. Past history of operations, hospitalization or blood transfusion.
3. Past anesthetic history with impact on previous airway problems during previous surgeries, hypersensitivity to anesthetic medications, any previous postoperative complications that could be attributed to anesthesia.
4. Family history for specific anesthetic problems like malignant hyperthermia.

B) Physical examination:

1- General examination. 2- Vital signs (heart rate, blood pressure, respiratory rate and temperature). 3- Heart, chest and abdominal examinations.

C) Anesthetic assessment:

1. Examination of the limbs for prediction of difficult cannulation.
2. Airway assessment.
3. Fasting hours: none of children were given any solid food 6 hours before the operation, but they were allowed to take clear fluids, soft drink or water until 2 hours before induction of anaeshesia.

D) Laboratory investigations:

1. Complete blood count (CBC).
2. Prothrombin time (PT), international normalized ratio (INR) and partial tissue thromboplastin time (PTT).

III- Demograghic data:

The patient's age, sex, weight, height and body mass index (BMI)were recorded.

IV-Intraoperative assessment:

1. Airway devices, anesthesia machine, ventilator, flowmeters and equipments were checked promptly.
2. Randomization: participants were randomly allocated to one of two equal groups, (group D) using orally given dexmedetomidine and (group MK) using orally given midazolam/ketamine using block randomization.

   Concealed allocation: closed envelope method for randomization containing code for dexmedetomidine group (D) or midazolam/ketamine group (MK). To ensure allocation concealment, the envelopes will be prepared by anesthesia nurse not involved in the study. Those enrolled after written informed consent were asked to pick one concealed envelope from the box and hand it over to the investigator concerned. The investigator then assigned to either (D) or (MK) according to the envelope code.

   Blinding: patients were blinded after assignment to interventions and randomly assigned into one of two equal groups. It was double blinded since the investigator was not aware of both groups.
3. During the preoperative visit, the researcher explained to the child and family what was done in the morning of surgery. The child was blinded to the used drug and was asked to choose a sealed envelope with his/her code number inside. The name, file number and body weight were recorded on the sealed envelope after been chosen. The on duty anesthetist was blinded to the premedication.
4. Parents were not aware of the premedication components, but oriented and agreed with our protocol. In the morning of operation, the study medications were prepared by a trained nurse into identical 10 ml syringes that were sequentially numbered. Each labeled syringe was mixed with apple juice to be given to the children. Premedication was given by one of the parents under supervision of anesthetist.
5. Premedication phase:The attending anesthetist in pre-anesthesia area reported the onset of premedication and level of sedation and the occurrence of vomiting was also monitored; children who vomited were excluded from the study. Thirty minutes after premedication, Parents accompanied their children till the Red-Line of the operating room, but their presence in the induction room was not be permitted according to the policy of the hospital.

Premedication was given orally to the children in the preanaesthetic room. (Group D) patients received dexmedetomidine(4 µg/kg) mixed with apple juice to fill the syringe up to 10 ml given orally and (group MK) patients received a combination of midazolam (0.5 mg/kg) and ketamine (1 mg/kg) mixed with apple juice to fill the syringe up to 10 ml and given orally.

Level of Sedation was assessed by Sedation Score (adapted from Wilton et al)(125)

Sedation and anxiolytics were evaluated in untouched patients. Then additional evaluation of cooperation e.g. (placement of the pulse oximetry sensor, electrocardiogram electrodes and mask induction of anesthesia) was performed.

The sedation score values were condensed to a variable consisting of three categories:

(Levels 1 and 2) Unacceptable conditions. (Levels 3 and 4) Acceptable conditions. (Level 5) Unacceptable deep sedation.

The behavior of the child during preoperative period was evaluated by the anesthesiologist using sedation score; the rating was performed at five different times:

(1) 2.5 minutes after oral drug administration. (2) 5 minutes after oral drug administration. (3)During separation from parents (at levels 3 and 4). (4) During introduction of the anesthesia mask to the child. (5) Immediately postoperative in PACU.

Whatever satisfaction of sedation was achieved or not after 60 min, anesthesia induction was performed.

Onset of sedation was defined as: the minimum time interval necessary for the child to become drowsy or asleep.

Peak sedative effect was defined as: the time interval from drug administration to reach the maximum level of sedation.

Both of onsets of sedation and peak sedative effect were recorded. Sedation and Anxiety levels were recorded every 15 min for a maximum time of 60 min after premedication In case a child came to the operating room already asleep, a steal induction was attempted.

Assessment of drug reaction after drug administration:

1=Crying 2=Not crying 3=Excessive salivation 4=Sneezing 5=cough

Evaluation of drug taste by 4-point scale after oral drug administration:

1. Good 3= Bitter
2. Indifferent 4= Unpleasant

6- Induction Phase: Children were transferred to the operating room; inhalational induction via transparent face mask (Jackson-Rees modification of Ayer's T-piece) was done using sevoflurane (Abbott, Abbott Park, Illinois, USA)started at a concentration of 1% and then increased every three breaths to a maximum of 8 % in 100% oxygen (6 L /min).The anesthetist asked the child to blow the balloon.

Five-point scale was used to assess Mask acceptance:

1. = Combative, crying
2. = Moderate fear of the mask, not easily calmed
3. = Cooperative with reassurance
4. = Calm, cooperative
5. = Asleep

   Mask induction scores of 1 and 2 were considered unsatisfactory. Scores of 3-5 were considered a successful response to premedication.

   After loss of consciousness, an intravenous line was inserted and when adequate depth of anesthesia was reached, endotracheal tube of appropriate size for the age and weight of the child was placed and patient was allowed to breathe spontaneously.

7- Intraoperative Monitoring: Monitoring equipment (Datex-Ohmeda, Helsinki, Finland™) was connected to each patient with standard monitoring including ECG, Non invasive blood pressure, Respiratory Rate, Pulse oximetry, Temperature and both inspiratory and end-expiratory Capnography.

Heart rate and blood pressure were recorded before premedication as a baseline then every 15 min until discharge.

8- Maintenance phase:

* The anesthetic was delivered in concentration that maintained a stable heart rate, blood pressure and respiratory rate (base line ±20%).
* Sevoflurane was reduced to 1.5-2 vol% in (30: 70%) oxygen and air ratio.
* Ventilation was assisted if the end-tidal carbon dioxide increased to ≥ 45 mmHg to be stabilized between 35-40 mmHg.
* At the end of procedure, anesthetic gas was discontinued and maintained on O2 100% > 5L/min
* Endotracheal tube was removed when the child showed adequate recovery from anesthesia; child was transferred to PACU for monitoring of vital signs till discharge to the ward.

At the end of anesthesia and before leaving operating room, assessment of recovery according to Modified Aldrete Recovery Score was done.

Adequate recovery was achieved if the score =10

9- Postoperative Period: Child was transferred to the post anesthesia care unit (PACU) for monitoring of vital signs till discharge to the ward.

In the PACU, parents were allowed to remain at the child's bedside immediately upon admission. A trained anesthesiologist, blinded to patient group assignment had been stayed with the patient until discharge to the ward.

Objective Pain Discomfort Score: was assessed, the intensity of pain immediately postoperatively, 30, 60 and 120 min thereafter (Objective Pain Discomfort Scale > 6 means pain and discomfort).

The parameters of this scale were:

Blood Pressure:

2 = > 20% preoperatively

1 = 11-20 % above preoperative 0 = < 11% preoperative

Crying:

2 =Crying not responding to TLC (Tender, Loving, Care)

1. = Crying but responds to TLC

0 = Not crying

Moving:

2 = Thrashing

1 = Restless 0 = None

Behavior:

2 = Hysterical

1 = Mild 0 = Patient asleep or calm

Verbal evaluation (language):

2 = Moderate pain (localizes verbally or pointing)

1 = Mild pain (cannot localize) 0 = Asleep or no pain

Assessment of agitation:

The state of agitation was assessed at arrival in the recovery room 30, 60 and 120 min postoperatively by means of a modified objective pain discomfort scale.

The modified objective pain Discomfort scale include movement, crying, and behavior items from the full OPS. For these three items, which constituted the modified OPS, the total possible score was 6.

Agitation was defined by a total score of ≥ 3 for these three items.

Patients were discharged when they were awake, had stable vital signs for at least 1 hour, had no pain or only mild pain, had not vomited for 1 hour, were able to tolerate clear fluid by mouth, and had no bleeding.

Duration of anaesthesia, duration of surgery, emergence time (time from the end of surgery till extubation) and recovery time (time from extubation till discharge from recovery): were recorded.

Time to the first request of postoperative analgesia: was recorded. The rescue analgesic was i.v.paracetamol at a dose of 15 mg/kg and if ineffective, fentanyl 0.5µg/kg bolus up to a total dose of 2µg/kg was used.

Complications of level of sedation (such as bradycardia, postoperative pain, shivering, PONV and emergence delirium): were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children with ASA I (American Society of Anesthesiologists physical status Grade I) = (normal healthy patients) or ASA II (American Society of Anesthesiologists physical status Grade II) = (patients with mild systemic disease and no functional limitations)
* Children scheduled for adenotonsillectomy

Exclusion Criteria:

* Children with central nervous system disorders & neurological problems.
* Children with inborn errors of metabolism.
* Obese children (BMI >30 kg/m2).
* Children with known allergy to dexmedetomidine, midazolam or ketamine.
* Children who vomit.
* Children with recent or chronic administration of sedative drugs, antipsychotics or tranquilizers.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Face mask acceptance | The anesthetist asked the child to blow the balloon for induction and assessment was recorded just after anesthesia induction
  Five-point scale was used to assess mask acceptance:
  1. = Combative, crying.
  2. = Moderate fear of the mask, not easily calmed.
  3. = Cooperative with reassurance.
  4. = Calm, cooperative.
  5. = Asleep, steal induction.
  (Scores 1 and 2): Unacceptable conditions. (Scores 3, 4 and 5): Acceptable conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elsadany, MD, Principal Investigator — Suez Canal University; Ghada Kamhawy, MD, Principal Investigator — Suez Canal University; Reda mohmd, MD, Principal Investigator — Suez Canal University; Mohamed Abdelgawad, MD, Study Director — Suez Canal University; Ahmed Elewa, MD, Principal Investigator — Suez Canal University
Locations (1):
- Anesthesia Department, Faculty of Medicine, Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No